CLINICAL TRIAL: NCT05260346
Title: Modulation of the Gut-brain Axis by Cranberries: Impact on University Students' Mental Wellbeing
Acronym: CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: The Cranberry Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CRANMOOD study
Record Dates: First submitted 2022-01-13; First posted 2022-03-02 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Cranberry flavored drink, once daily, in a 8fl oz bottle. Identical in appearance and taste compared with the treatment.
  Interventions: Dietary Supplement: Placebo
- Cranberry juice (Active Comparator): 100% cranberry juice, once daily, in a 8fl oz bottle.
  Interventions: Dietary Supplement: Cranberry juice

INTERVENTIONS:
Dietary Supplement: Cranberry juice — composition: Water, cranberry juice concentrate
  Arms: Cranberry juice
Dietary Supplement: Placebo — composition: Water, dextrose, citric acid, malic acid, fumaric acid, colorants, xanthan gum, natural flavor, emulsion
  Arms: Placebo

SUMMARY:
In this work, the investigators will assess whether cranberry (poly)phenols improve mood disorders including stress, anxiety and depression via the gut-brain axis in university students. The investigators will evaluate whether the effects observed are related to an improvement in gut microbiome diversity and function, and whether the mechanism of action may be mediated by a decrease in inflammatory markers, modulation of neurotransmitters or via an alteration of BDNF levels. The investigators will also quantify the most comprehensive panel of cranberry (poly)phenol metabolites. A double-blind, randomized placebo controlled 2-arm parallel study will be conducted in the Metabolic Research Unit (MRU, Department of Nutritional Sciences at KCL).

DETAILED DESCRIPTION:
The study population will be final year BSc and MSc university students between 20-25 years old (n=60), who are generally healthy and not taking any medication. The study will be conducted during the period prior to their final exams (January until September). The intervention will be cranberry and placebo juice, consumed daily for 12 weeks, and will be provided free of cost by the Cranberry Institute. After a screening visit to evaluate inclusion and exclusion criteria, informed consent will be obtained, and subjects will be randomized to the treatments.

The study will consist in a total of 4 visits, one visit every 4 weeks over a total of 12 weeks intervention. Volunteers will consume a cranberry or a control drink every day for 12 weeks. The day before each visit (pre-visit), volunteers will self-collect a total of 6 saliva samples throughout the day to measure cortisol levels as a biomarker of stress. Mental health, cognitive function, diet and physical activity will also be assessed using self-reported questionnaires, an online cognitive battery test and an online 24 h dietary recall. In addition, on the day before visits 1 and 4 (baseline and 12 weeks), a stool sample will be self-collected to assess changes in gut microbiome diversity and composition. On the day of each visit, a spot urine sample will be self-collected after waking up and before breakfast. During each visit, volunteers will drop the self-collected samples, and will collect new kits for the next visit. Visits 1 and 4 will last approximately 20 min, while visits 2 and 3 will last approximately 5 minutes. In addition, during visits 1 and 4, blood samples will be taken to investigate changes in gut-brain axis and cranberry related metabolites. Blood samples will also be collected at baseline to assess general health status of participants (blood lipids, markers of liver and kidney function, urea, uric acid, creatinine, and glucose).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 20-25 years old.
* Final year BSc or MSc university students.
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study.
* Able to understand the nature of the study.
* Able and willing to give signed written informed consent.
* Comply with all study protocol procedures.

Exclusion Criteria:

* Subjects taking regular prescribed medication (including iron for anemia).
* Grade 1 hypertensive or above, as defined as SBP superior or equal to 140 mmHg or DBP superior or equal to 90 mmHg.
* Obese participants, defined as BMI superior or equal to 30.
* Diabetes mellitus and metabolic syndrome.
* Chronic and acute disease.
* Terminal renal failure and other kidney abnormalities.
* Malignancies.
* Allergies to berries or other significant food allergy.
* Subjects who took food supplements, dietary supplement or herbal remedies within 1 month of study start.
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet.
* Subjects with allergies to berries or other relevant/related food.
* Subjects who reported participant in another study within one month before the study start.
* Subjects who smoke an irregular number of cigarettes per day or plan quitting smoking in the next 3 months.
* Subjects who require chronic antimicrobial or antiviral treatment
* Subjects with unstable psychological condition (diagnosed with mental health disorders).
* Subjects with history of cancer, myocardial infarction, cerebrovascular incident
* Pregnant, lactating or planning to become pregnant, as well as pre-menopausal women who do not have a regular menstrual cycle and do not adequate method of contraception.
* Any reason or condition that in the judgement of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Changes in mood | Baseline and 12 weeks
  Mood measured as the Total Mood Disturbance (TMD), using the Profile of Mood States (POMS) questionnaire. The POMS assessment has six scales of measure: Anger-Hostility, Confusion-Bewilderment, Depression-Dejection, Fatigue-Inertia, Tension-Anxiety, and Vigor-Activity. Scores on these items are added together to determine a Total Mood Disturbance score. Additionally, there is a measure of Friendliness which is scored separately. The POMS2 is an adjective checklist with instructions to respond "How have you been feeling over the PAST WEEK, INCLUDING TODAY" on a 5- point Likert response scale ranging from 0 = Not at all to 4 = Extremely. If one changes the instructions to "how you feel RIGHT NOW" then the instrument measures emotional states. This it is adaptable to both state and trait forms of affect. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Mental Health outcomes: stress levels | Baseline and 12 weeks
  Mental Health outcomes including changes in stress levels, measured as salivary and blood cortisol and the Perceived Stress Scale (PSS) questionnaire. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. It consists of 10 questions, takes 5-10 minutes to complete and is for individual or group administration. Higher scores indicate higher levels of perceived stress.
Mental Health outcomes: anxiety | Baseline and 12 weeks
  Mental Health outcomes including changes in anxiety and depression symptoms, measured with the Hospital Anxiety and Depression Scale (HADS) questionnaire. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. For both scales (anxiety and depression), higher scores mean a worse outcome.
Changes in cognitive function and performance | Baseline and 12 weeks
  Measured using the Online General Cognitive Assessment Battery (CogniFit) using established procedures. The cognitive score is an aggregate measure of the current cognitive strength of different cognitive skills. The minimum cognitive score is 0 and the maximum is 800. A higher score means higher cognitive abilities.
Changes in plasma gut-brain-axis metabolites | Baseline and 12 weeks
  Serotonin and kynurenine pathway will be measured using targeted metabolomics
Changes in brain-derived neurotrophic factor | Baseline and 12 weeks
  Brain-derived neurotrophic factor (BDNF) will be measured using established procedures
Changes in inflammatory markers | Baseline and 12 weeks
  Inflammatory markers, including blood cytokines (IL1β, IL2, IL4, IL6, IL8, IL10, IL12, IL13, MIF, IFN-γ, and TNF-α), will be measured using established procedures
Changes in plasma and faecal short chain fatty acids | Baseline and 12 weeks
  Measured using gas chromatography according to established procedures
Changes in plasma and urinary cranberry polyphenol metabolites | Baseline and 12 weeks
  Measured using a validated targeted metabolomics method
Assessment of habitual diet | Baseline and 12 weeks
  Diet will be assessed using 7-day food diaries (from the European Prospective Investigation into Cancer and Nutrition) at baseline and after 12 weeks.
Assessment of physical activity | Baseline and 12 weeks
  The international physical activity questionnaire (IPAQ) will also be used to assess physical activity. IPAQ assesses physical activity undertaken across a comprehensive set of domains including leisure time, domestic and gardening (yard) activities, work-related and transport-related activity. The higher the score, the higher the physical activity level.
Changes in gut microbiome diversity and composition. | Baseline and 12 weeks
  Faecal samples will be collected at baseline and 12 weeks after consumption of cranberry or placebo drinks. Gut microbiome diversity and composition will be analysed using 16s mRNA sequencing at the Genome Centre of Queen Mary University (London, UK).

OTHER OUTCOMES:
Changes in plasma metabolome | Baseline and 12 weeks
  Measured via untargeted metabolomics using liquid chromatography mass spectrometry
Changes in urinary metabolome | Baseline and 12 weeks
  Measured via untargeted metabolomics using liquid chromatography mass spectrometry
Changes in gene expression | Baseline and 12 weeks
  Measured using microarray hybridization and data analyses on Affymetrix CEL files using GeneSpring GX software
Changes in DNA methylation | Baseline and 12 weeks
  Measured using the Illumina Infinium HD Methylation Assay
Changes in blood pressure | Baseline and 12 weeks
  Blood pressure measured as systolic and diastolic blood pressure after 12-week daily consumption of cranberry
Changes in sleep patterns | Baseline and 12 weeks
  Measured as bedtime and sleep duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No